CLINICAL TRIAL: NCT03601260
Title: To Examine the Percentage of Cases of Acute Treatment With Allopurinol in Gout Patients as Secondary Treatment
Brief Title: The Percentage of Cases of Acute Treatment With Allopurinol in Gout Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-FKH-1
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gout Patients (Other): Allopurinol 100 mg-300mg/day as secondary treatment in gout patients
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Treatment of gout patients by oral dosage of 100 mg-300mg/ day of Allopurinol

SUMMARY:
The aim of the study is to determine the percentage of cases of acute treatment with Allopurinol in gout patients who have been previously treated.

ELIGIBILITY:
Inclusion Criteria:

* Gout patients

Exclusion Criteria:

* Pregnant women
* Chronic renal failure
* Patients with Allopurinal hypersensitivity

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Gout patients treated with Allopurinol | Six months
  Retrospective identification through medical records of percentage of gout patients treated with Allopurinol

SECONDARY OUTCOMES:
Patients with contraindication to Allopurinol | Six months
  Retrospective identification through medical records of percentage of gout patients with contraindications to Allopurinol

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No